CLINICAL TRIAL: NCT03589248
Title: Predictive Value of Transabdominal Intestine Sonography in Critically Ill Patients：A Prospective, Observational Study
Brief Title: Predictive Value of Transabdominal Intestine Sonography in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, research assistant, Nanjing PLA General Hospital
Other Study IDs: 2016NLYZDRC015
Record Dates: First submitted 2018-06-23; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Gastrointestinal Dysfunction; Critical Illness; Intestine Ultrasonography
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GIF score: assess the AGI by gastrointestinal failure(GIF) score
  Interventions: Diagnostic Test: GIF score; Diagnostic Test: US score
- US score: assess the AGI by ultrasonography(US) score
  Interventions: Diagnostic Test: GIF score; Diagnostic Test: US score

INTERVENTIONS:
Diagnostic Test: GIF score — assessment by GIF score
Diagnostic Test: US score — assessment by ultrasonography score

SUMMARY:
It is very important to evaluate the degree of gastrointestinal dysfunction in critical ill patients. Thus the investigators conducted transabdominal intestine ultrasonography(US) in critical ill patients to evaluated the degree of gastrointestinal dysfunction under the acute gastrointestinal injury (AGI)

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years
* Acute Physiology Chronic Health Evaluation II (APACHE II) score >8

Exclusion Criteria:

* uncontrolled mesenteric vascular disease
* uncontrolled chronic organ dysfunction
* advanced cancer
* any terminal stage disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe complications after surgery and severe trauma
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
predict value of 28-day mortality | one and a half year
  predict value of 28-day mortality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao T, Cheng MH, Xi FC, Chen Y, Cao C, Su T, Li WQ, Yu WK. Predictive value of transabdominal intestinal sonography in critically ill patients: a prospective observational study. Crit Care. 2019 Nov 27;23(1):378. doi: 10.1186/s13054-019-2645-9. PMID 31775838